CLINICAL TRIAL: NCT04846036
Title: A Randomized Placebo Controlled, Double-blind Phase II Study to Explore the Safety, Efficacy and Pharmacokinetics of Sonlicromanol in Children With Genetically Confirmed Mitochondrial Disease
Brief Title: The KHENERGYC Study
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic company decision - not related to safety concerns
Sponsor: Khondrion BV (Industry)
Collaborators: Julius Clinical (Industry); ProPharma Group (Industry); Europees Fonds voor Regionale Ontwikkeling (EFRO) (Unknown); Ardena (Unknown); Certara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH176-204
Record Dates: First submitted 2021-02-05; First posted 2021-04-15 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-05

CONDITIONS: Mitochondrial Diseases; Mitochondrial DNA tRNALeu(UUR) m.3243A<G Mutation; MELAS; Subacute Necrotizing Encephalomyelopathy
Keywords: KH176; Sonlicromanol; MELAS; Leigh syndrome; Oxidative phosphorylation (oxphos); Phase II
MeSH Terms: conditions — Mitochondrial Diseases; MELAS Syndrome; Leigh Disease | interventions — 6-hydroxy-2,5,7,8-tetramethylchroman-2-carboxylic acid

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonlicromanol (Experimental): Paediatric-equivalent dose (as determined by Physiologically Based Pharmacokinetics (PBPK) modelling and the results of the Adaptive PK study) of sonlicromanol twice daily administered as an oral liquid for 26 weeks
  Interventions: Drug: Sonlicromanol
- Placebo (Placebo Comparator): Matching placebo twice daily orally for 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sonlicromanol — Oral administration of sonlicromanol twice daily
  Other Names: KH176
  Arms: Sonlicromanol
Drug: Placebo — Oral administration of matching placebo twice daily
  Arms: Placebo

SUMMARY:
This a randomized placebo controlled, double-blind phase II study to explore the pharmacokinetics, safety and efficacy of sonlicromanol in children (from birth to 17 years) with genetically confirmed mitochondrial disease of which the gene defect is known to decrease one or more oxidative phosphorylation system enzymes and who suffer from motor symptoms ("KHENERGYC").

DETAILED DESCRIPTION:
Mitochondrial Diseases (MD) are rare progressive, multi-system, often early onset and fatal disorders affecting both children and adults. Despite advances in the understanding of mitochondrial disorders, treatment options are extremely limited and, to date, largely supportive. Therefore, there is an urgent need for novel treatments. Sonlicromanol (KH176) is an orally bio-available small molecule under development for the treatment of these disorders. The current study will explore the pharmacokinetics, safety and efficacy of sonlicromanol in children (from birth to 17 years) with genetically confirmed mitochondrial disease of which the gene defect is known to decrease one or more oxidative phosphorylation system enzymes and who suffer from motor symptoms.

The primary objective of the study is to evaluate the effect of sonlicromanol on motor symptom severity in children with genetically confirmed mitochondrial disease affecting oxidative phosphorylation during a 6 month treatment period (GMFM).

The trial consists of 2 phases, with the main phase being a randomized placebo controlled, double-blind, phase II parallel group study to explore the efficacy and safety of sonlicromanol in twenty-four (24) children with mitochondrial disease and motor symptoms,.

The first phase is an adaptive PharmacoKinetics (PK) study with 4 days treatment (to expected steady state in most subjects) in the following age-groups: birth - 1 year, 1-2 years, 2- 6 years, 6-12 years, and 12 - 17 years. An age group should have at least 3 subjects before being analysed. Subjects will take 4 days of open-label sonlicromanol orally at the anticipated adult-equivalent dose. After completion of enrolment in an age group, the PK data from that age group will be analysed to confirm the adult-equivalent dose that will be used thereafter in the second phase of the trial. Older age groups will be studied before younger age groups.

In the second phase subjects will be randomized (by age group) over 2 groups. Group 1 will receive an adult-equivalent dose of sonlicromanol twice daily orally for 26 weeks. Group 2 will receive matching placebo twice daily for 26 weeks. A final follow-up visit is scheduled 2 weeks after the intake of the last dose of the treatment period.

Duration of Subject Participation:

The overall study duration of the trial for a eligible subject is estimated to be approximately 7 months, consisting of up to 4 weeks screening, 26 weeks (6 months) of treatment and 2 week post-treatment follow-up. At the end of the study treatment all participants will be offered to continue treatment with sonlicromanol during a open label extension (OLE) trial for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 0 months and 17 years
2. Genetically confirmed mitochondrial disease, of which the gene defect is known to decrease one or more oxidative phosphorylation system enzymes and who suffer from motor symptoms, based on investigator judgement
3. Abnormal gross motor function and/or presence of at least one clinically significant motor symptom (hypotonia, decreased muscle strength, ataxia, dystonia, chorea and/or spasticity) based on investigator judgement
4. Before enrollment in the adaptive PK phase and before randomization into the double-blind placebo-controlled phase: Gross Motor Function Measure-88 (GMFM-88) Total Score ≤96%
5. Before enrollment in the adaptive PK phase and before randomization into the double-blind placebo-controlled phase: International Paediatric Mitochondrial Disease Scale IPMDS Score ≥10
6. Stable disease symptoms since the previous routine control visit (consistent with a score of "stable" on the item "disease course since previous IPMDS" of the IPMDS) in the opinion of the investigator.
7. Written informed (patient/parental/caregiver) consent, able and willing to comply with the study requirements of the study protocol.
8. Women of childbearing potential must be willing to use highly effective contraceptive methods during the entire study, i.e. combined (estrogen and progestogen containing) oral, intravaginal or transdermal hormonal contraception associated with inhibition of ovulation; oral, injectable, or or implantable progestogen-only hormonal contraception associated with inhibition of ovulation; use of an intrauterine device; an intrauterine hormone releasing system, bilateral tubal occlusion and vasectomy of the partner. Any hormonal contraception method must be supplemented with a barrier method (preferably male condom). Vasectomised partner is considered a highly effective birth control method provided that partner is the sole sexual partner of the subject and that the vasectomised partner has received medical assessment of the surgical success. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. Reliability of sexual abstinence needs to be evaluated in in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Note 1: Natural family planning methods, female condom, cervical cap or diaphragm are not considered adequate contraceptive methods in the context of this study.

Note 2: To be considered not of childbearing potential, potential female subjects must have been surgically sterilized (bilateral tubal ligation, hysterectomy or bilateral oophorectomy) for at least 6 months prior to Screening.

Note 3: KH176 has been shown non-genotoxic judged from the Ames test, Chromosomal Aberration test and in vivo Micronucleus test. Moreover, appreciable systemic exposure from the exposure to (~2.5 mL) semen is extremely unlikely. However, until reproductive toxicology studies have confirmed that KH176 does not adversely affect normal reproduction in adult males and females, as well as causing developmental toxicity in the offspring, the following contraceptive precautions must be adhered to:

* male subjects with female partners of childbearing potential must be willing to use condoms during the entire study.
* female partners of childbearing potential of male subjects must be willing to use adequate contraceptive methods during the entire study, i.e., a hormonal contraceptive method (pill, vaginal ring, patch, implant, injectable, hormone-medicated intrauterine device) or an intrauterine device.

Exclusion criteria:

1. Surgery of the gastro-intestinal tract with removal of piece(s) of stomach, duodenum or jejunum that might interfere with absorption. Feeding through gastrostomy tube is however allowed.
2. Treatment with an investigational product within 3 months or 5 times the half-life of the investigational product (whichever is longer) prior to the first dose of the study medication.
3. Clinically relevant cardiovascular disease or risk factors for arrythmia:

   1. Abnormal ECG (including QTcF exceeding the 95th percentile for the age- and sex-dependent QTc interval (https://www.qtcalculator.org) and/or abnormal structural or functional 2D ECHO
   2. Systolic Blood Pressure (SBP) above the 95th percentile for the sex, age group and height percentile at screening or baseline on single measurement (see appendix 1)
   3. History of acute or chronic heart failure, (family) history of unexplained syncope or congenital long and short QT syndrome or sudden death
   4. Hyperkalemia or hypokalemia; hypomagnesemia or hypermagnesemia; hypocalcemia or hypercalcemia (local laboratory normal values; to be judged by investigator)
4. Clinically relevant abnormal laboratory results:

   1. Aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) > 3 times upper limit of normal (ULN), or bilirubin > 3 x ULN. If a patient has ASAT or ALAT > 3 x ULN but < 3.5 x ULN, re-assessment is allowed at the investigator's discretion.
   2. Estimated glomerular filtration rate below age-appropriate limits (according to the formula: 40.9* ((1.8 / Cystatine C)0.93):

      < 2 months: < 25 ml/min/1.73 m2 2 months to 1 year: < 35 ml/min/1.73 m2 > 1 year: < 60 ml/min/1.73 m2
   3. All other clinically relevant parameters at screening or baseline as judged by the investigator
5. History of hypersensitivity or idiosyncrasy to any of the components of the investigational product.
6. Medical history of drug abuse (illegal drugs such as cannabinoids, amphetamines, cocaine, opiates or problematic use of prescription drugs such as benzodiazepines, opiates).
7. The use of any of the following medication and/or supplements within 4 weeks or 5 times the half-life (whichever is longer) prior to the first dosing of the study medication:

   1. (multi)vitamins, co-enzyme Q10, Vitamin E, riboflavin, and antioxidant supplements (including, but not limited to idebenone/EPI-743, mitoQ); unless stable for at least one month before first dosing and remaining stable throughout the study.
   2. any medication negatively influencing mitochondrial functioning (including but not limited to valproic acid, glitazones, statins, anti-virals, amiodarone, and non-steroidal anti- inflammatory drugs (NSAIDs)), unless stable for at least one month before first dosing and remaining stable throughout the study.

      Note: thus, mitoQ and any medication negatively influencing mitochondrial functioning are allowed as long as the dose has been stable for at least one month prior to first dosing and remains stable throughout the study.
   3. any strong Cytochrome P450 (CYP)3A4 inhibitors (all 'conazoles-anti-fungals', HIV antivirals, grapefruit).
   4. strong CYP3A4 inducers (including HIV antivirals, carbamazepine, phenobarbital, phenytoin, rifampicin, St. John's wort, pioglitazone, troglitazone).
   5. any medication known to affect cardiac repolarisation, unless the QTc interval at screening is normal during stable treatment for a period of two weeks, or 5 half-lives of the medication and its major metabolite(s), whichever period is the shortest (all anti-psychotics, several anti-depressants: nor- / amitriptyline, fluoxetine, anti-emetics: domperidone (Motilium®), granisetron, ondansetron).
   6. any medication metabolised by CYP3A4 with a narrow therapeutic width.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Motor Symptom Severity as assessed with the Gross Motor Function Measure-88 (GMFM-88) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the GMFM-88.The GMFM-88 consists of 88 questions and assesses motor function in 5 domains (lying and rolling; sitting; crawling and kneeling; standing; walking, running, and jumping). 4-point scoring system for each item, item scores ranges from 0-3. Higher scores denote better performance. Scaled score indicates the percentage of total score. Total score ranges from 0-100%

SECONDARY OUTCOMES:
Fine manual motor skills as assessed with the 9 Hole Peg Test (NHPT) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the NHPT. The NHPT examines the fine hand motor skills by assessing the speed of movement of the hand.The fastest time of 2 attempts is recorded for the dominant hand as well as the non-dominant hand. When the maximum time is reached (50 seconds) the number of transported rods is counted (maximum = 18; minimum = 0). Faster times (in sec) and higher number of rods denote better performance.
Spasticity as assessed with the Modified Tardieu Scale for spasticity (MTS) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the MTS. The MTS quantifies spasticity by assessing the muscle's response to stretch applied at three specified velocities (as slow as possible; speed of limb falling under gravity; moving as fast as possible) and rating the intensity and duration of the muscle reaction to stretch and the joint angle. The quality of the muscle reaction (spasticity grade) is scored on a 5-grade scale (range: 'No resistance throughout the course of the movement' to 'Joint immovable'). Lower scores denote better performance. The Spasticity Angle X is the difference between the angles of arrest at slow speed and of catch-and release or clonus at fast speed; the Spasticity Grade Y is an ordinal variable that grades the intensity (gain) of the muscle reaction to fast stretch. The outcome parameter of angle (in degrees, range: 0-180 degrees) can only be determined with spasticity grade 2 and higher.
Dystonia as assessed with Dystonia (Barry-Albright Dystonia scale (BAD) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the BAD. The BAD assesses dystonia in eight body regions: eyes, mouth, neck, trunk, and the four extremities. Dystonia is scored as none (0), slight (1), mild (2), moderate (3), or severe (4). Individual scores for each region are added for a total score. total score ranging from 0-32. A higher score denotes worse outcome.
Ataxia as assessed with the Scale for the Assessment and Rating of Ataxia (SARA) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the SARA. The SARA is a semi- quantitative assessment of a range of different impairments in cerebellar ataxia. The scale is an 8-item based scale related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test. The score ranges from 'no ataxia' (0) to 'most severe ataxia' (40). A higher score denotes worse outcome.
Disability as assessed with the PEDI-CAT (Paediatric Evaluation of Disability Inventory (PEDI-CAT) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the PEDI-CAT. The PEDI-CAT is a computer adaptive caregiver report which estimates a child's abilities from a minimal number of the most relevant items or from a set number of items within three functional domains: Daily Activities, Mobility, Social/Cognitive, and Responsibility. <= 30 items per domain. Higher scores denote better performance.
Mitochondrial disease signs and symptoms as assessed with the International Paediatric Mitochondrial Disease Scale (IPMDS) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the IPMDS. The IPMDS assesses all aspects of mitochondrial disease by exploring three domains: a) 'complaints and symptoms' (23 items), b) 'physical examination' (21 items) and c) 'functional tests' (13 items). The domain and total scores are expressed as the percentage of items which were feasible to perform (maximum = 100%; minimum = 0%. A higher score denotes better performance.
Caregiver burden as assessed with the ZARIT-12 Burden scale (ZBI-12) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the ZBI-12. The ZBI-12 assesses caregiver perceptions of burden by indicating the extent of burden experienced while providing care to their child. The responses on the scale range from 'not at all' to 'extremely'. Total scores are obtained by summing the item scores, maximum = 48; minimum = 0). higher scores denote higher burden.
Quality of life as assessed with the Neurology Quality of life short Form (NeuroQL-SF) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the NeuroQL-SF. The Fatigue Short Form Paediatric version is an 8-item score evaluating the perception of fatigue and its impact in daily life activities. Scores on individual items range from 1-5. The total score ranges from 5-40. Higher score denotes worse outcome.
Clinician-scored global impression of change (CGIC) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the CGIC. The CGIC assesses the clinician's perception of the degree to which patient's illness/symptoms have improved or worsened following intervention using a 7-point Likert scale. Score ranges from 1-7. A higher score denotes worsening of symptoms.
Patient/Caregiver scored global impression of change (PGIC) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the PGIC. The PGIC assesses patient's/caregiver's perception of the degree to which patient's illness/symptoms have improved or worsened following intervention using a 7-point Likert scale. Score ranges from 1-7. A higher score denotes worsening of symptoms.
Patient/Caregiver scored impression of change on patient-identified 3 Most Bothersome Symptoms (MBSA) caused by mitochondrial disease | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the MBSA. The MBSA assesses patient/caregiver scored impression of the degree to which each of the 3 patient-identified most bothersome symptoms caused by mitochondrial disease have improved or worsened following intervention. Score ranges from 1-7 for each of the symptoms. A higher score denotes worsening of symptoms.
Growth as assessed by weight | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of weight in kilogram (Kg)
Growth as assessed by height | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of height in centimeters (cm)
Growth as assessed by head circumference | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of head circumference in centimeters (cm), for children younger than 3 years only.
Growth as assessed by Body Mass Index (BMI) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of BMI, weight and height will be combined to report BMI in kg/m^2 children aged 3 years and above
Temperature | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of temperature in degree Celsius
10 meter Walk Test (10MWT) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the 10MWT. The 10MWT assesses the patients' physical ability to walk/run, the patients' walking speed and stamina. The patient is instructed to walk/run 10 meters and the time is measured while the patient walks the set distance. Faster times (in sec) denotes better performance.

OTHER OUTCOMES:
Mortality | Up to 29 weeks
  Mortality rate during treatment
Health Utility Index (HUI) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the HUI. The HUI is measuring health status and health-related quality of life (HRQL) on multiple dimensions of health status, including vision, hearing, speech, ambulation/mobility, pain, dexterity, self-care, emotion and cognition and a HRQL score for overall health. Each dimension has 3- 6 levels. Overall HRQL scores range from 0.00 to 1.00. A higher score denotes better quality of life/health.
EQ-5D-Y Proxy | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the EQ-5D-Y. The EQ-5D-5L-Y (proxy 1) measures health in five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 response categories (levels): no problems, slight problems, moderate problems, severe problems and extreme problems. The patient's health state is indicated in a 1-digit number expressing the level selected for that dimension. The digits for the five dimensions are combined into a 5-digit number that describes the patient's health state, ranging from 11111 (having no problems in all dimensions) to 55555 (having extreme problems in all dimensions). A higher score denotes a worse health state.
EQ-Visual Analogue Scale (EQ-VAS) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of the EQ-VAS.The EQ-VAS measures perceived health, ranging from 0 ('The worst health you can imagine') to 100 ('The best health you can imagine'). Range: 0-100, a higher score denotes better health.
Overall survival | Up to 29 weeks
  Overall survival over 29 weeks
Palatability of sonlicromanol as assessed with the five level Facial Hedonic Scale (FHS) and Visual Analogue Scale (VAS) | Day 1
  FHS combined with a 100-point linear visual analogue scale (VAS), with point 0 aligning with the extreme left of the facial prompt used in the FHS and point 100 aligning with the extreme right side of the FHS. The score ranges from 0 -100. A higher score denotes a better outcome/higher palatability.
Acceptability of sonlicromanol as assessed by patient/caregiver daily reporting of acceptability. | Up to 27 weeks
  The acceptability of sonlicromanol is determined by daily assessment of acceptability by reporting if the subject has 'swallowed the total dose', 'spat out (part of) the dose', or 'refused to take dose'. Total acceptability scores are obtained by summing the number of doses totally swallowed, spat out or refused.
HbA1c: mmol Glycated Hb per mol Hb | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment of HbA1c. Glucose homeostasis / diabetes control
Electrocardiogram (ECG): PQ interval (milliseconds) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Mean and the maximum change from baseline to each assessment in PQ interval.
Electrocardiogram (ECG): QRS duration (milliseconds) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Mean and the maximum change from baseline to each assessment in QRS duration.
Electrocardiogram (ECG): T peak - T end interval | Baseline (Day 1), week 6, week 13, week 27, week 29
  Mean and the maximum change from baseline to each assessment in T peak - T end interval.
Electrocardiogram (ECG): QTc | Baseline (Day 1), week 6, week 13, week 27, week 29
  Mean and the maximum change from baseline to each assessment in QTc.
Electrocardiogram (ECG): T wave morphology: peak, symmetry | Baseline (Day 1), week 6, week 13, week 27, week 29
  Mean and the maximum change from baseline to each assessment in T wave morphology: peak, symmetry.
Treatment Emergent Adverse Events (TEAEs) | up to 29 weeks
  Frequency of TEAEs throughout the study period
Systolic Blood Pressure (mmHG) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in systolic blood pressure (mmHG)
Diastolic Blood Pressure (mmHG) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in diastolic blood pressure (mmHG)
Heartrate (Beats Per Minute (BPM)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment Heartrate in beats per minute (BPM)
Haematology: Concentration of haemoglobin (Hb) in mmol/L | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in haemoglobin (Hb) concentration in mmol/L
Haematology: Haematocrit (Ht): Volume of RBC as fraction of total blood volume (L/L). | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in haematocrit (Ht) in L/L
Haematology: Mean Corpuscular Haemoglobin (MCH) in pg/cell (average mass of Hemoglobin (Hb) per red blood cell (RBC)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in mean corpuscular haemoglobin (MCH) in pg/cell
Haematology: Concentration of Mean Corpuscular Haemoglobin Concentration (MCHC) (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in mean corpuscular haemoglobin concentration in mmol/L
Haematology: Red Blood Cell Count (RBC) (cell/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in Red Blood Cell (RBC) count in cells/L
Haematology: MCV Mean Corpuscular Volume of ared blood cells in femtoliter (fL) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in mean corpuscular volume (MCV) of red blood cells in fL
Haematology: White Blood Cell (WBC) count (cells/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in white blood cell (WBC) count (cells/L)
Haematology: white blood cell differential (WBC differential: neutrophils, lymphocytes, monocytes, eosinophils, basophils) count (cells/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in WBC differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils) count in cells/L
Haematology: Thrombocytes count (cells/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in thrombocytes count in cells/L
Haematology: Total protein (g/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in total protein in g/L
Chemistry: Concentration of Alkaline Phosphatase (Units/L (U/L)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in alkaline phosphatase concentration in U/L
Chemistry: Concentration of Aspartate Aminotransferase (ASAT) (Units/L (U/L)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in aspartate aminotransferase (ASAT) concentration in U/L
Chemistry: Concentration of Alanine Aminotransferase (ALAT) (Units/L (U/L)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in Alanine Aminotransferase (ALAT) concentration in U/L
Chemistry: Concentration of gamma-Glutamyl Transferase (gamma-GT) (Units/L (U/L)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in gamma-Glutamyl Transferase (gamma-GT) concentration in U/L
Chemistry: Concentration of total bilirubin (umol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in total bilirubin concentration in umol/L)
Chemistry: Concentration of urea (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in urea concentration in mmol/L
Chemistry: Concentration of creatinine (umol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in creatinine concentration in umol/L
Chemistry: Concentration of creatinine kinase (Units/L (U/L)) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in creatinine kinase concentration in U/L
Chemistry: Concentration of sodium (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in sodium concentration in mmol/L
Chemistry: Concentration of potassium (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in potassium concentration in mmol/L
Chemistry: Concentration of calcium (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in calcium concentration in mmol/L
Chemistry: Concentration of chloride (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in chloride concentration in mmol/L
Chemistry: Concentration of lactate (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in lactate concentration in mmol/L
Chemistry: Concentration of Thyroid-stimulating Hormone (TSH) (mE/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in Thyroid-stimulating Hormone concentration in mE/L
Chemistry: Concentration of free Thyroxine (fT4) (pmol/l) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment visit in free Thyroxine (fT4) concentration in pmol/L
Chemistry: Concentration of C-reactive protein (CRP) (mg/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in C-reactive protein (CRP) concentration in mg/L
Chemistry: Concentration of lipase (U/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in lipase concentration in U/L
Chemistry: Concentration of uric acid (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in uric acid concentration in mmol/L
Chemistry: Concentration of phosphate (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in phosphate concentration in mmol/L
Chemistry: Concentration of human serum albumin (g/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in human serum albumin concentration in g/L
Chemistry: Concentration of glucose (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in glucose concentration in mmol/L
Chemistry: Concentration of Lipids: cholesterol, triglycerides, low density lipoproteins (LDL), high density lipoproteins (HDL) (mmol/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in Lipids concentration: cholesterol, triglycerides, low density lipoproteins (LDL), high density lipoproteins (HDL) in mmol/L
Chemistry: Concentration of amylase (U/L) | Baseline (Day 1), week 6, week 13, week 27, week 29
  Changes from baseline to each assessment in amylase concentration in U/L
Metabolomics: Concentration of Fibroblast Growth factor 15 (FGF-15) (pg/mL) | Baseline (Day 1), week 27
  Changes from baseline to each assessment in FGF-15 concentration in pg/mL)
Metabolomics: Concentration of Growth Differentiation Factor-15 (GDF-15) (pg/mL) | Baseline (Day 1), week 27
  Changes from baseline to each assessment in GDF-21 concentration (in pg/mL)
Pharmacokinetics: Time-to-peak drug plasma concentration (Tmax) (hours) | Baseline (Day 1), Week 27
  Tmax: Time to reach maximum (peak) plasma concentration following drug administration (hours)
Pharmacokinetics: Peak drug concentration (Cmax) (ng/mL) | Baseline (Day1), week 27
  Changes from baseline to week 27 in Tmax: Maximum (peak) plasma drug concentration in ng/mL
Pharmacokinetics: Ctrough (ng/mL) | Baseline (Day1), week 27
  Changes from baseline to week 27 in plasma concentration (measured concentration at the end of a dosing interval at steady state in ng/mL
Pharmacokinetics: AUCinf (h*ng/mL) | Baseline (Day1), week 27
  Changes from baseline to week 27i n Area under the plasma concentration time curve from time zero to infinity in h*ng/mL
Pharmacokinetics: AUCtau (h*ng/mL) | Baseline (Day1), week 27
  Changes from baseline to week 27 in Area under the plasma concentration time curve in h*ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Lonneke de Boer, MD, Principal Investigator — Radboud University Medical Center Nijmegen, Netherlands
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smeitink J, van Maanen R, de Boer L, Ruiterkamp G, Renkema H. A randomised placebo-controlled, double-blind phase II study to explore the safety, efficacy, and pharmacokinetics of sonlicromanol in children with genetically confirmed mitochondrial disease and motor symptoms ("KHENERGYC"). BMC Neurol. 2022 Apr 27;22(1):158. doi: 10.1186/s12883-022-02685-3. PMID 35477351